CLINICAL TRIAL: NCT04341818
Title: Vitamin D and Resistance Exercise in Elderly
Brief Title: Vitamin D and Resistance Exercise in Elderly (NUTRIAGINGVitD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Karl-Heinz Wagner, Professor of Human Nutrition, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FA219002_2
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Aging
Keywords: aging; vitamin D; resistance training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strength Training and Vitamin D monthly (Experimental): Four weeks of Vitamin D (50.000 IU once per month) followed by a 10 week guided resistance training (progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the vitamin D intake remains. Over the whole study period participants get 400 mg calcium/day.
  Interventions: Other: Strength Training and Vitamin D monthly
- Strength Training and Vitamin D daily (Experimental): Four weeks of Vitamin D (800 IU once per day) followed by a 10 week guided resistance training (progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the vitamin D intake remains. Over the whole study period participants get 400 mg calcium/day.
  Interventions: Other: Strength Training and Vitamin D daily
- Strength Training and no Vitamin D (Experimental): Four weeks of no vitamin D administration followed by a 10 week guided resistance training (progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the vitamin D intake remains. Over the whole study period participants get 400 mg calcium/day.
  Interventions: Other: Strength Training and no Vitamin D

INTERVENTIONS:
Other: Strength Training and Vitamin D monthly — For 4 wks 50.000 IU vitamin D is given as a monthly dose together with daily 400mg of calcium. Both as a supplement, followed by a 10 weeks resistance training (progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the vitamin D and calcium intake remain.
  Arms: Strength Training and Vitamin D monthly
Other: Strength Training and Vitamin D daily — For 4 wks 800 IU vitamin D is given as a daily dose together with daily 400mg of calcium. Both as a supplement, followed by a 10 weeks resistance training (progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the vitamin D and calcium intake remain.
  Arms: Strength Training and Vitamin D daily
Other: Strength Training and no Vitamin D — For 4 wks no vitamin D is administered, followed by a 10 weeks resistance training (progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the also no vitamin D is given. Over the whole study period participants get 400 mg calcium/day.
  Arms: Strength Training and no Vitamin D

SUMMARY:
The aim of this randomized, double-blind, controlled intervention study with parallel groups is to investigate the effect of resistance training (2x/week for 10 weeks) with and without different goals of vitamin D intake on muscle strength, function and mass, oxidative stress parameters and the immune system in community dwelling persons. Participants (n = 100) will be community-dwelling older adults. After a preparticipation screening and a vitamin D blood investigation (vitamin D status below 75 nmol/L) participants will be distributed randomly but stratified by sex, age and initial vitamin D plasma levels to one of the 3 groups (Vitamin D daily + strength training, Vitamin D monthly + strength training, no Vitamin D + strength training).

Study participants are eligible if they are male or female with an age between 65 and 85 years and if their cognitive status as well as their physical fitness level allows to participate at the strength training sessions. Exclusion criteria comprise chronic diseases which contraindicate the training sessions, serious cardiovascular disease, diabetic retinopathy and manifest osteoporosis, a frailty index at or above 3, medication with anticoagulants or cortisone drugs, a regular strength training during the last six months and a vitamin D plasma concentration of 75nmol/L or above.

Primary outcome measure is the change in the handgrip strength. Secondary outcome measures comprise anthropometric data, functional performance tests, immunological and oxidative stress parameters, DNA/Chromosomal damage microbiota, metabolomics and the nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the age of 65 and 85 years
* Adequate mental condition in order to follow the instructions and to perform the resistance exercise independently (Mini-Mental-State >23)
* Independently mobile

Exclusion Criteria:

* Chronic diseases, which contraindicate a training participation
* Serious cardiovascular diseases (congestive chronic heart failure, severe or symptomatic aortic stenosis, unstable angina pectoris, untreated arterial hypertension, cardiac arrhythmias)
* Diabetic retinopathy
* Manifest osteoporosis
* Regular use of cortisone-containing drugs
* Regular strength training (> 1x / week) in the last 6 months before inclusion
* Vitamin D plasma level of 75 nmol/l or above

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in handgrip strength (kg) | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  Handgrip strength of the right hand will be measured to the nearest kilogram (kg) using a hand Dynamometer. Participants will be encouraged to perform a maximal contraction within approximately 4 to 5 s. After a rest of 60 s, participants will be asked to perform a second trial. The highest score of maximum voluntary contraction will be used for data analyses.

SECONDARY OUTCOMES:
Change from baseline in chair stand test (repetitions within 30s) | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  The maximum number of completed cycles of unsupported chair rises (from a seated to a fully erected position (hip and knees straightened)) completed within 30 s is counted automatically (Leonardo Mechanography). Force, acceleration, power, kinetic energy, potential energy, mass, total duration, time per iteration are reported as secondary parameters.
Change from baseline in muscle mass with BIA (kg) | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
Change from baseline in 6min walking test (distance in meter) | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  Participants are instructed to walk alone as quickly as possible (without running) around a 30 m shuttle course as many times as possible within the time limit of 6 mins.
Change from baseline in the composition of gut-microbiota | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  Gene sequencing of the 16S rRNA on the stool samples are performed to identify the microbes down to genus level as well as the microbial diversity and relative abundance.
Change from baseline in stool short-chain fatty acids (SCFAs) | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  The stool short-chain fatty acids (SCFAs) will be extracted and quantitatively analysed by gas chromatography.
Change from baseline in oxidative stress marker such as malondialdehyde | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  The investigators will consider changes in plasma concentrations of oxidative stress marker such as malondialdehyde.
Change from baseline in inflammatory marker (i.g. IL-6, TNF-alpha) | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  The investigators will consider changes in plasma concentrations of Interleukin 1 (IL-1), IL-6, IL-8, IL-10, TNF-alpha
Change from baseline in the metabolomic response | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  The metabolomic response (ie all metabolites) to the interventions will be analyzed using both nuclear magnetic resonance (NMR) and mass spectrometry (MS) techniques. Patterns of metabolites will be evaluated with statistical techniques, ie discriminant analysis and principal component analysis.
Change from baseline in the amino acid pattern | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  The plasma amino acid pattern will be assessed with HPLC-MS.
Change from baseline in DNA damage (%DNA in the tail) | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  DNA damage will be assessed in lymphocytes, whole blood and urine in response to the interventions.
Change from baseline in chromosomal damage (number of micronuclei/1000 binucleated cells) | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  Chromosomal damage will be assessed in lymphocytes in response to the interventions.
Change from baseline in RDA and DNA gene expression | baseline, after dietary intervention (4 weeks) and after dietary intervention and strength training (14 weeks)
  RNA and DNA gene expression will be assessed in response to the interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided